CLINICAL TRIAL: NCT02771665
Title: Mammographic Density and the Risk of Tumor Recurrence in Asian Women: a Case-control Study
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401068RIND
Record Dates: First submitted 2016-05-11; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Case Control Study

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Breast cancer women with known recurrences: Breast cancer women with known recurrences (locoregional recurrence and distant metastasis)
  Interventions: Other: Mammographic breast density at diagnosis
- Breast cancer women without recurrences: Breast cancer women without recurrences
  Interventions: Other: Mammographic breast density at diagnosis

INTERVENTIONS:
Other: Mammographic breast density at diagnosis — Mammographic breast density at diagnosis

SUMMARY:
To evaluate the influence of mammographic breast density at diagnosis on the risk of cancer recurrence and survival outcome in patients with invasive breast cancer after surgery

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with invasive breast cancer between 2004 and 2009 who had undergone surgery and had the mammographic breast density ascertained before, or at, diagnosis.

Exclusion Criteria:

* Women diagnosed with invasive breast cancer between 2004 and 2009 who had not undergone surgery or who had no mammographic breast density ascertained before, or at, diagnosis.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with invasive breast cancer who had undergone surgery between 2004 and 2009
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Hazard ratios for recurrence | 2004 to 2009

SECONDARY OUTCOMES:
Hazard ratios for death | 2004 to 2009

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Ling-Yu Chen, MD, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang YS, Chen JL, Huang CS, Kuo SH, Jaw FS, Tseng YH, Ko WC, Chang YC. High mammographic breast density predicts locoregional recurrence after modified radical mastectomy for invasive breast cancer: a case-control study. Breast Cancer Res. 2016 Dec 1;18(1):120. doi: 10.1186/s13058-016-0784-3. PMID 27906044